CLINICAL TRIAL: NCT02564991
Title: Cross-Sectional and Longitudinal Study of Structural Imaging
Brief Title: Study of Structural Imaging
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150203; 15-AA-0203
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Chemically-Induced Disorders; Substance-Related Disorders; Mental Disorders; Alcohol Dependence; Alcohol-Related Disorders
Keywords: Alcoholism; MRI; Structural MRI; Cerebellum; Natural History
MeSH Terms: conditions — Chemically-Induced Disorders; Substance-Related Disorders; Mental Disorders; Alcoholism; Alcohol-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: 125 non-substance abusing controls (NSAC)
- Individuals with Alcohol Use Disorder: This group includes individuals who enrolled NIAAA alcohol treatment.

SUMMARY:
Background:

The way alcohol affects brain structure has been widely studied. But the way it affects all parts of the brain is still unknown. Researchers want to use magnetic resonance imaging (MRI) scans to study brain structure and function. They hope this will help them better understand changes that happen in brain regions during treatment of alcohol use disorders.

Objectives:

To study changes in the brain by using MRI in people with and without alcohol use disorders. To study how brain changes affect gait, balance, cognitive ability, and behavior. To see how the brain recovers when alcohol use stops.

Eligibility:

People with alcohol dependence who are currently hospitalized in a particular unit at NIH.

Healthy volunteers 30 60 years old without an alcohol use disorder.

Design:

Participants will be screened under a separate protocol.

Participants will give a urine sample for a drug test and pregnancy test at each study visit. They will also have to pass a breath alcohol test.

At the first visit, participants will have an MRI. The scanner is a metal cylinder in a strong magnetic field. Participants will lie on a table that slides in and out of the cylinder.

They will do behavior and memory tasks outside the scanner.

They will have gait and balance tested. They will have to stand on both legs, stand on just one leg, and walk in a straight line. They will perform each task with eyes open, then with eyes closed.

They will have tests of memory, thinking, and problem solving.

Some participants will have a second visit. They will have another MRI and repeat some of the behavior and memory tasks.

...

DETAILED DESCRIPTION:
Objective

The purpose of this protocol is to characterize cerebellar volumes and function in alcoholics and recovery of cerebellar volume and function during early abstinence. This study also investigates how cerebrocerebellar circuits contribute to cognitive and motor impairment in alcoholism.

Study Population

Healthy volunteers and Inpatient participants with alcohol use disorders.

Design

Participants will receive whole-brain structural imaging and assessment of cerebellar function at the time of admission and again at the time of discharge.

Outcome

The Primary outcome of this study is to assess recovery of cerebellar structure and function at the end of treatment compared to treatment entry measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 30 to 60 years old
  2. Physically healthy
  3. Healthy volunteers only: Currently consuming 7 or less standard drinks per week if female; 14 or less drinks per week if male.

EXCLUSION CRITERIA:

1. Significant history of head trauma or cranial surgery,
2. History of diabetes or stroke which requires medical intervention,
3. Clinical or laboratory evidence of severe hepatic disease as determined by ALT or AST greater than 5 times the upper normal limit, INR greater than 2.0, total bilirubin greater than 2.5 mg/dL, and albumin lower than 3.0 g/dL.
4. Positive HIV test.
5. Healthy volunteers only: 5 or more binge drinking episodes in the past 30 days (5 or more standard drinks on one occasion for males, 4 or more standard drinks on one occasion for females within two hours)
6. Healthy volunteers only:

   --Have fulfilled DSM-IV or DSM-5 criteria for current alcohol use disorder or substance abuse disorder
7. Inpatient participants only: Currently experiencing symptoms of withdrawal from alcohol (As determined by the most recent measurement within the past 30 days CIWA score > 8)
8. Female participants only: Are currently pregnant
9. IPresence of any contraindication for fMRI as determined by the NIAAA MRI Safety Screening Questionnaire
10. Have calustrophobia

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy volunteers and Inpatient participants with alcohol use disorders. . Design Participants will receive whole-brain structural imaging and assessment of cerebellar function at the time of admission and again at the time of discharge
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
The Primary outcome of this study is to assess recovery of cerebellar structure and function at the end of treatment compared to treatment entry measures. | Entry and End of Treatment
  To assess recovery of cerebellar structure and function at the end oftreatment compared to treatment entry measures.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Momenan, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-AA-0203.html